CLINICAL TRIAL: NCT04067960
Title: Precision Pharmacogenomics in Cancer Patients
Brief Title: Pharmacogenomics Testing in the Optimal Use of Supportive Care Medications in Stage III-IV Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19-002006; NCI-2019-04725 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-002006 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Biliary Tract Carcinoma; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Malignant Brain Neoplasm; Malignant Genitourinary System Neoplasm; Malignant Solid Neoplasm; Pancreatobiliary Carcinoma; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Pancreatic Cancer; Stage IVA Prostate Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Pancreatic Cancer; Stage IVB Prostate Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Brain Neoplasms; Urogenital Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — Specimen Handling; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (pharmacogenomics testing) (Experimental): Patients undergo one-time collection of saliva sample for pharmacogenomics testing. Patients also complete quality of life assessment at baseline and at 3 months after pharmacogenomics testing.
  Interventions: Procedure: Biospecimen Collection; Other: Genetic Testing; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of saliva
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Genetic Testing — Undergo pharmacogenomics testing
  Other Names: genetic analysis; Genetic Examination; Genetic Test
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial studies how well a genetic test called pharmacogenomics works in directing the optimal use of supportive care medications in patients with stage III-IV cancer. Pharmacogenomics is the study of how genes may affect the body's response to and interaction with some prescription medications. Genes, which are inherited from parents, carry information that determines things such as eye color and blood type. Genes can also influence how patients process and respond to medications. Depending on the genetic makeup, some medications may work faster or slower or produce more or fewer side effects. Pharmacogenomics testing may help doctors learn more about how patients break down and process specific medications based on their genes and improve the quality of life of cancer patients receiving clinical care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate patient perceptions surrounding their quality of life (QOL) prior to pharmacogenomics (PGx) testing and 3 months post PGx testing.

II. Understand the clinical utility/relevancy of PGx testing in cancer patients at Mayo Clinic Arizona from the viewpoint of their providers.

OUTLINE:

Patients undergo one-time collection of saliva sample for pharmacogenomics testing. Patients also complete quality of life assessment at baseline and at 3 months after pharmacogenomics testing.

After completion of study, patients are followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patient enrolled to Mayo Clinic IRB: 18-000326
* Patients with stage 3 or 4 breast, colorectal, prostate/genitourinary (GU), pancreato-biliary, brain, melanoma, and ovarian cancer
* Individuals have agreed to participate and signed the study informed consent form

Exclusion Criteria:

* Patients with cancer types other than the ones mentioned above
* Patient with psychiatric illness, or situations that would limit compliance with the study requirements or the ability to willingly give written informed consent
* Previous PGx testing with results available within Mayo Clinic electronic medical record (EMR)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Changes in symptoms, quality of life (QOL), and perceptions about pharmacogenomics (PGx) testing | Baseline up to 3 months post consent
  Patient survey responses will be compared across administration time points to look for changes in symptoms, QOL, and perceptions about PGx testing.

SECONDARY OUTCOMES:
Provider opinions surrounding the clinical utility/relevancy of PGx testing in cancer patients | Up to 3 months
  Will qualitatively assess provider opinions surrounding the clinical utility/relevancy of PGx testing in cancer patients via the provider survey. Provider survey responses will be examined to determine the range of perceptions and experiences associated with PGx testing and result reporting for patient tests. Descriptive statistics will be used to report provider survey results.

CONTACTS AND LOCATIONS:
Overall Officials: Jewel Samadder, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States